CLINICAL TRIAL: NCT02482311
Title: A Phase Ib, Open-Label, Multi-Centre Study to Assess the Safety, Tolerability, Pharmacokinetics, and Anti-tumour Activity of AZD1775 Monotherapy in Patients With Advanced Solid Tumours
Brief Title: Safety, Tolerance, PK, and Anti-tumour Activity of AZD1775 Monotherapy in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6015C00001; REFMAL 383 (Other: SCRI Development Innovations, LLC)
Record Dates: First submitted 2015-06-11; First posted 2015-06-26 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Cancer, TNBC, SCLC, Other Solid Tumours
Keywords: AZD1775; Ovarian cancer (BRCA1/2 mutation); Ovarian cancer (PARP-failure); Triple negative breast cancer (TNBC); Small-cell lung cancer (SCLC); Solid tumours
MeSH Terms: conditions — Ovarian Neoplasms; Triple Negative Breast Neoplasms; Small Cell Lung Carcinoma | interventions — adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD1775 (Experimental): Single-arm study. AZD1775 will be administered for 3 consecutive days at the start of week 1 and week 2 of each 21-day cycle.
  This study will be conducted in two parts, designated Part A and Part B. Part A is a safety lead-in. Part B will commence after the safety lead-in and will investigate the safety and efficacy of AZD1775 monotherapy in expansion cohorts of specific tumour types.
  Interventions: Drug: AZD 1775

INTERVENTIONS:
Drug: AZD 1775 — AZD1775 will be taken orally approximately every 12 hours over 3 days at the start of week 1 and week 2 of each 21-day cycle (Days 1-3 and 8-10), for a total of 12 doses with each treatment cycle.
  AZD1775 should be taken approximately 2 hours before or 2 hours after food.

SUMMARY:
This is an open-label, multi-centre, Phase Ib study of AZD1775 designed to assess the safety, tolerability, pharmacokinetics, and anti-tumour activity of AZD1775 monotherapy in patients with advanced solid tumours.

DETAILED DESCRIPTION:
This study is being conducted in two parts, designated Parts A and B. Part A is a safety lead-in consisting of a cohort of approximately 12 patients with advanced solid tumours.

Part B expansion cohorts will investigate AZD1775 monotherapy in advanced tumour types with molecular biomarkers of interest. The tumour types to be evaluated are: 1) ovarian cancer (BRCA1/2 mutation [PARP-failures]), 2) ovarian cancer (BRCA wild-type) with more than three prior lines of treatment, 3) triple negative breast cancer (TNBC), and 4) small-cell lung cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Previous chemotherapy for recurrent or metastatic disease.
3. Measurable disease is required for Part B expansion cohorts according to RECIST v1.1 criteria.
4. Radiation therapy completed at least 7 days prior to start of study treatment and patients must have recovered from any acute adverse effects.
5. ECOG Performance Status (PS) score of 0-1.
6. Baseline laboratory values as follows:

   1. ANC ≥1500/μL
   2. Hgb ≥9 g/dL
   3. Platelets ≥100,000/μL
   4. ALT and AST ≤3 x ULN or ≤5 x ULN if known hepatic metastases.
   5. Serum bilirubin WNL or ≤1.5 x the ULN in patients with liver metastases; or total bilirubin ≤3.0 x ULN with direct bilirubin WNL in patients with well documented Gilbert's Syndrome.
   6. Serum creatinine ≤1.5 x the ULN and a calculated creatinine clearance (CrCl) ≥45 mL/min by the Cockcroft-Gault method.
7. Negative serum or urine pregnancy test within 3 days prior to start of study treatment.
8. Fertile male patients willing to use at least one medically acceptable form of birth control for the duration of the study and for 2 weeks after treatment stops.
9. Predicted life expectancy ≥12 weeks.

Inclusion Criteria Specific for Part A:

1. Histologically or cytologically documented, locally advanced or metastatic solid tumour, excluding lymphoma, for which standard therapy does not exist or has proven ineffective or intolerable.
2. Has agreed to the collection of archival tumour tissue or recent tumour biopsy tissue, it taken for routine clinical purposes at baseline if archival tissue is not available, for molecular biomarker analyses.

Inclusion Criteria Specific for Part B:

1. Ovarian cancer defined as a histologically confirmed diagnosis of epithelial ovarian, fallopian tube, or primary peritoneal cancer refractory to standard therapies of for which no standard therapy exists. Confirmed BRCA1 or BRCA2 mutation from a prior test. Patient progressed while receiving and/or following treatment with a PARP-inhibitor for advanced disease (recurrent or metastatic.
2. Ovarian cancer confirmed BRCA wild-type from a prior test.
3. Triple-negative breast cancer (TNBC) defined as histologically confirmed diagnosis of breast cancer and must have received at least 1 chemotherapy-containing regimen for advanced disease (recurrent or metastatic). Tumour must be triple-negative, defined as minimal or no expression of estrogen and progesterone receptors [<10% of cells positive by immunohistochemistry (IHC)], and minimal or no expression of HER2 (IHC staining 0 or 1+ or FISH-).
4. Small-cell lung cancer (SCLC) defined as a histologically confirmed diagnosis of SCLC and must have received at least 1 chemotherapy-containing regimen for advanced disease (recurrent or metastatic).

Exclusion Criteria:

1. Any chemotherapy within 3 weeks of the first dose of AZD1775, except hormonal therapy in the refractory cohort.
2. Use of a study drug ≤21 days or 5 half-lives, whichever is shorter.
3. Major surgical procedures ≤28 days, or minor procedures ≤7 days.
4. Grade >1 toxicity from prior therapy (except alopecia or anorexia).
5. CNS disease other than neurologically stable, treated brain metastases.
6. Prescription or non-prescription drugs or other products known to be sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued two weeks prior to Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study drug.
7. NYHA ≥ Class 2.
8. Mean resting corrected QT interval (QTc) ≥450 msec for males and ≥470 msec for females.
9. Pregnant or lactating.
10. Serious active infection, or serious underlying medical condition.

12. Presence of other active invasive cancers. 13. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs), serious adverse events (SAEs) and dose-limiting toxicities (DLTs) as a measure of safety and tolerability. | From first dose of study treatment up to last day of Cycle 1 (21 days)
  The AZD1775 dose is considered safe and tolerable if ≤ 1 of 6 patients experiences a DLT.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Every 6 weeks until treatment discontinuation as defined by RECIST 1.1, projected 12 months.
  The proportion of patients achieving a complete or partial tumour response (CR or PR) according to RECIST 1.1 criteria.
Disease Control Rate (DCR) | Every 6 weeks until treatment discontinuation as defined by RECIST 1.1, projected 12 months
  The proportion of patients achieving a complete response (CR) or partial response (PR), or stable disease (SD) according to RECIST v1.1 criteria
Duration of Response (DoR) | Every 6 weeks until treatment discontinuation as defined by RECIST 1.1, projected 12 months
  The time from first documented tumor response until the date of documented progression or death from any cause.
Progression Free Survival (PFS) | Every 6 weeks until treatment discontinuation as defined by RECIST 1.1, project 12 months.
  Defined as the time from date of first dose of AZD1775 until the date of objective disease progression or death by any cause as defined by RECIST 1.1.
PK profile: Plasma concentrations of AZD1775 and PK parameters (Cmax, C8hr, tmax, AUC, tlast, t½λz) | Pre-dose and 1, 2, 4, 6, 8 and 12 hours post-dose of AZD1775 during Cycle 1-Day 1 and Cycle 1-Day3 or Day-10 of the safety lead-in part of study
  Blood samples will be collected at various timepoints post-dosing
QTc prolongation | ECGs collected pre-dose and 1, 2, 4, 6, 8 and 12 hours post-dose in Cycle 1-Day 1 and on Cycle 1-Day 3 or Day 10.
  ECGs will be obtained at various timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Todd M. Bauer, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (16):
- United States (13):
  - Research Site, Fayetteville, Arkansas
  - Research Site, San Francisco, California
  - Research Site, West Hollywood, California
  - Research Site, Fort Myers, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Detroit, Michigan
  - Research Site, Charlotte, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Milwaukee, Wisconsin
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario

REFERENCES:
- [Derived] Bauer TM, Moore KN, Rader JS, Simpkins F, Mita AC, Beck JT, Hart L, Chu Q, Oza A, Tinker AV, Imedio ER, Kumar S, Mugundu G, Jenkins S, Chmielecki J, Jones S, Spigel D, Fu S. A Phase Ib Study Assessing the Safety, Tolerability, and Efficacy of the First-in-Class Wee1 Inhibitor Adavosertib (AZD1775) as Monotherapy in Patients with Advanced Solid Tumors. Target Oncol. 2023 Jul;18(4):517-530. doi: 10.1007/s11523-023-00965-7. Epub 2023 Jun 6. PMID 37278879
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6015C00001&attachmentIdentifier=023dd524-b5bd-49b9-afe2-ee168fff47de&fileName=D6015C00001_CSP_Redacted.pdf&versionIdentifier=